CLINICAL TRIAL: NCT05512949
Title: A Phase 2 Randomized, Open-Label, Multisite Trial to Evaluate the Immunogenicity of Dose Reduction Strategies of the MVA-BN Vaccine
Brief Title: Trial to Evaluate the Immunogenicity of Dose Reduction Strategies of the MVA-BN Monkeypox Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0020A
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2022-08-23

CONDITIONS: Monkeypox
Keywords: Dose Reduction; Immunogenicity; JYNNEOS; Monkeypox; MVA-BN; Open-Label; Randomized; Vaccine
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): 0.1 mL of 2 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29. N=70
  Interventions: Biological: JYNNEOS
- Arm 2 (Experimental): 0.05 mL of 1 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29. N=70
  Interventions: Biological: JYNNEOS
- Arm 3 (Active Comparator): 0.5 mL of 1 x 10^8 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered subcutaneously on Days 1 and 29. N=70
  Interventions: Biological: JYNNEOS

INTERVENTIONS:
Biological: JYNNEOS — JYNNEOS is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. Each 0.5 mL dose is formulated to contain 0.5 x 10^8 to 3.95 x 10^8 infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Subcutaneous is administered in the deltoid region, intradermal is administered in the volar aspect (inner side) of the forearm.

SUMMARY:
This study is a Phase 2 randomized, open-label, non-placebo controlled, multi-site clinical trial that will evaluate two intradermal (ID) regimens for Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) vaccine compared to the standard subcutaneous (SC) regimen in healthy, vaccinia-naïve adults 18 to 50 years of age, inclusive. At least 210 participants will be enrolled and randomized to one of three study arms. The two dose sparing strategies include one-fifth (2 x 10^7) and one-tenth (1 x 10^7) of the standard dose of MVA-BN administered ID on Day 1 and 29 (Arm 1 and 2, respectively). The comparator arm (Arm 3) will be the 2-dose standard (1 x 10^8) MVA-BN SC regimen.

The study will enroll a 1:1:1 randomization allocation. Participants will not be stratified by clinical trial site, demographic characteristics or human immunodeficiency virus (HIV) infection status; however, these data will be collected during screening and enrollment. Each participant may be screened either in a separate visit in the 7 days prior to Day 1 or on Day 1.

The primary hypothesis involves a two-step hierarchical process. The study will first test non-inferiority of the 2 x 10^7 ID regimen relative to 1 x 10^8 SC (standard dose regimen). If the 2 x 10^7 ID regimen is non-inferior to the standard dose regimen, hypothesis testing will proceed to test non-inferiority of the 1 x 10^7 ID regimen relative to the standard dose regimen.

The primary objectives are: 1) to determine if peak humoral immune responses following an ID regimen of 2 x 10^7 50% Tissue Culture Infectious Dose (TCID50) MVA-BN are non-inferior to the licensed regimen of 1 x 10^8 MVA-BN administered SC; 2) to determine if peak humoral immune responses following an ID regimen of 1 x 10^7 TCID50 MVA-BN are non-inferior to the licensed regimen of 1 x 10^8 MVA-BN administered SC.

DETAILED DESCRIPTION:
This study is a Phase 2 randomized, open-label, non-placebo controlled, multi-site clinical trial that will evaluate two intradermal (ID) regimens for Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) vaccine compared to the standard subcutaneous (SC) regimen. This study will enroll healthy, non-pregnant, non-breastfeeding adults 18 to 50 years old inclusive. Participants with stable medical conditions and well-controlled human immunodeficiency virus (HIV) infection can participate. At least 210 participants will be enrolled and randomized to one of three study arms. The two dose sparing strategies include one-fifth (2 x 10^7) and one-tenth (1 x 10^7) of the standard dose of MVA-BN administered ID on Day 1 and 29 (Arm 1 and 2, respectively). The comparator arm (Arm 3) will be the 2-dose standard (1 x 10^8) MVA-BN SC regimen.

The study will enroll a 1:1:1 randomization allocation. Participants will not be stratified by clinical trial site, demographic characteristics or HIV infection status; however, these data will be collected during screening and enrollment. Each participant may be screened either in a separate visit in the 7 days prior to Day 1 or on Day 1.

The primary hypothesis involves a two-step hierarchical process. The study will first test non-inferiority of the 2 x 10^7 ID regimen relative to 1 x 10^8 SC (standard dose regimen). If the 2 x 10^7 ID regimen is non-inferior to the standard dose regimen, hypothesis testing will proceed to test non-inferiority of the 1 x 10^7 ID regimen relative to the standard dose regimen.

The primary objectives are: 1) to determine if peak humoral immune responses following an ID regimen of 2 x 10^7 50% Tissue Culture Infectious Dose (TCID50) MVA-BN are non-inferior to the licensed regimen of 1 x 10^8 MVA-BN administered SC; 2) to determine if peak humoral immune responses following an ID regimen of 1 x 10^7 TCID50 MVA-BN are non-inferior to the licensed regimen of 1 x 10^8 MVA-BN administered SC.

The secondary objectives are: 1) to determine if individual peak humoral immune responses following each ID regimen are non-inferior to the licensed regimen administered SC; 2) to evaluate humoral immune responses of each ID regimen (separately) compared to licensed SC regimen each study day; 3) to evaluate the kinetics of the humoral immune responses of each ID regimen (separately) compared to licensed SC regimen through Day 365; 4) To compare relative safety among study arms as assessed by systemic and local reactogenicity for 14 days after each vaccination, unsolicited adverse events for 28 days after each vaccination, and serious adverse events (SAE) and medically attended events (MAAE) from Day 1 through Day 57, and related SAE/MAAEs through Day 181.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18 - 50 years of age inclusive at the time of consent.
2. Able to read the written informed consent, states willingness to comply with all study procedures, and is anticipated to be available for all study visits.
3. Agreement to adhere to Lifestyle Considerations during the study.
4. Females of reproductive potential who have sexual intercourse with males must agree to use highly effective contraception for at least 1 month prior to signing ICF and through Day 57.
5. In good general health as evidenced by medical history, physical examination, and clinical judgement of the investigator to be in stable state of health.

   *Participants with pre-existing stable chronic medical conditions defined as conditions not requiring significant change in therapy or hospitalization for worsening disease in the 4 weeks prior to enrollment can be included at the discretion of the investigator. This includes stable, well-controlled HIV positive individuals.
6. If HIV infected individual, they must be on suppressive Antiretroviral therapy (ART) for at least 6 months, report a cluster of differentiation 4 (CD4) count of greater than 350 cells/uL and no Acquired Immune Deficiency Syndrome (AIDS)-defining illness in the last year.

Exclusion Criteria:

1. Ever received a licensed or an investigational smallpox or monkeypox vaccine.

   *This includes Dryvax, Acam2000, LC 16 m8, Modified Vaccinia Ankara (MVA)-based vaccine candidate or licensed vaccines, and Jynneos, Imvamune or Imvanex).
2. Any history of monkeypox, cowpox, or vaccinia infection.
3. Close contact of anyone known to have monkeypox in the 3 weeks prior to signing Informed Consent Form (ICF).
4. Immunocompromised as determined by the investigator.
5. Recent or current use of any immunosuppressing medications in the 4 weeks prior to signing ICF.

   **Topical, ophthalmic, inhaled, intranasal and intraarticular corticosteroids are acceptable, but receipt of >/= 20 mg/day of prednisone or equivalent for >/= 14 consecutive days in the 4 weeks prior to signing ICF is exclusionary.
6. Pregnant or breast feeding.
7. Received or plans to receive a live vaccine in the 4 weeks prior to signing ICF and 4 weeks after each vaccination.
8. Received or plans to receive any other vaccine in the 2 weeks prior to signing ICF through Day 43.
9. Received experimental therapeutic agent or vaccine in the 3 months prior to signing ICF.
10. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products.

    ***This includes individuals with history of severe allergic reaction to gentamicin, ciprofloxacin, chicken or egg protein.
11. Has tattoos, scars, or other marks which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
12. Has any medical disease or condition that, in the opinion of the participating site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.

    * This includes acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, San Diego (UCSD) - Antiviral Research Center (AVRC), San Diego, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - The Hope Clinic of Emory University, Decatur, Georgia
  - NIH Clinical Research Center, Investigational Drug Management and Research Section, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Frey SE, Baden LR, El Sahly HM, Davey RT, Rebolledo PA, Diemert DJ, Little SJ, Creech CB, Oikonomopoulou Z, Sherman AC, Whitaker JA, Rouphael NG, Desrosiers A, Martin TCS, Rolsma SL, Hoet B, Watanabe A, Jaunarajs A, Moss B, Tomashek KM, Lerner A, Beigel JH; DMID 22-0020 Study Group. Evaluation of the safety and immunogenicity of two fractional intradermal regimens of MVA-BN compared to standard dose vaccination. Vaccine. 2026 Jan 1;69:127959. doi: 10.1016/j.vaccine.2025.127959. Epub 2025 Nov 29. PMID 41319397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy, non-pregnant, non-breastfeeding adults 18 to 50 years old recruited from the communities at large surrounding 8 clinical sites throughout the U.S. The enrollment period occurred between 09SEP2022 and 12OCT2022.
Groups:
- 2 x 10^7 ID MVA-BN: 0.1 mL of 2 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29.
  JYNNEOS: JYNNEOS is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. Each 0.5 mL dose is formulated to contain 0.5 x 10^8 to 3.95 x 10^8 infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Intradermal vaccination is administered in the volar aspect (inner side) of the forearm.
- 1 x 10^7 ID MVA-BN: 0.05 mL of 1 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29.
  JYNNEOS: JYNNEOS is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. Each 0.5 mL dose is formulated to contain 0.5 x 10^8 to 3.95 x 10^8 infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Intradermal vaccination is administered in the volar aspect (inner side) of the forearm.
- 1 x 10^8 SC MVA-BN: 0.5 mL of 1 x 10^8 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered subcutaneously on Days 1 and 29.
  JYNNEOS: JYNNEOS is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. Each 0.5 mL dose is formulated to contain 0.5 x 10^8 to 3.95 x 10^8 infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Subcutaneous vaccination is administered in the deltoid region.
Period: Overall Study
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Started | 75 | 78 | 76
Completed | 69 | 68 | 71
Not Completed | 6 | 10 | 5
Not completed — Lost to Follow-up | 4 | 6 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Completion status unknown | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 x 10^7 ID MVA-BN: 0.1 mL of 2 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29.
- 1 x 10^7 ID MVA-BN: 0.05 mL of 1 x 10^7 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered intradermally on Days 1 and 29.
- 1 x 10^8 SC MVA-BN: 0.5 mL of 1 x 10^8 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered subcutaneously on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN | Total
Number analyzed (Participants) | 75 | 78 | 76 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 78 | 76 | 229
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (8.9) | 31.6 (8.9) | 32.7 (9.1) | 32.2 (8.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender Man | 40 | 36 | 36 | 112
  Cisgender Woman | 29 | 41 | 37 | 107
  Genderqueer | 1 | 0 | 0 | 1
  Gender Non-binary | 3 | 1 | 1 | 5
  Gender Non-conforming | 0 | 0 | 1 | 1
  Transgender Man/Trans Man | 1 | 0 | 0 | 1
  Transgender Woman/Trans Woman | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0
  Decline to state | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 37 | 112
  Male | 42 | 36 | 39 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 22 | 47
  Not Hispanic or Latino | 65 | 63 | 54 | 182
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 11 | 9 | 7 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 13 | 14 | 38
  White | 50 | 51 | 47 | 148
  More than one race | 2 | 4 | 4 | 10
  Unknown or Not Reported | 1 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 75 | 78 | 76 | 229
HIV Status [Count of Participants; unit: Participants]
  HIV Negative | 73 | 75 | 73 | 221
  HIV Positive | 2 | 3 | 3 | 8
Sexual Identity [Count of Participants; unit: Participants]
  Heterosexual or straight | 46 | 54 | 48 | 148
  Lesbian or gay | 11 | 10 | 19 | 40
  Bisexual | 13 | 8 | 6 | 27
  Queer | 2 | 3 | 1 | 6
  Pansexual | 1 | 2 | 0 | 3
  Asexual | 2 | 1 | 1 | 4
  Other | 0 | 0 | 0 | 0
  Decline to state | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Vaccinia Virus Specific Plaque Reduction Neutralization Test (PRNT) Geometric Mean Titer (GMT) at Day 43
Description: Venous blood was collected at Study Day 43 and the serum was analyzed via the PRNT assay to determine if GMT of the intradermal regimen of 2 x 10^7 TCID50 MVA-BN and 1 x 10^7 TCID50 MVA- BN were non-inferior to that of the licensed regimen of 1 x 10^8 TCID50 MVA-BN administered subcutaneously.
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood sample for immunogenicity testing for which valid results were reported. Participants are analyzed according to the study product that they received.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 74 | 75 | 76
titer | 203.2 [164.5 to 250.9] | 113.2 [90.3 to 141.9] | 288.9 [222.4 to 375.2]
Statistical Analysis 1: Comparison: 2 x 10^7 ID MVA-BN vs 1 x 10^8 SC MVA-BN; The selection of the noninferiority (NI) margin was based on the pivotal Phase 3 trial by Pittman et al., in 2019 comparing one dose of ACAM2000 and the now licensed 2-dose standard MVA-BN regimen, which provided an estimated relative (peak) immune response of approximately 2-times higher for MVA-BN. An NI margin of 0.5 corresponds to an immune response of the lower-dose MVA-BN at least as high as what would be expected for ACAM2000; Test type: Non-Inferiority — The ID-dose regimen is considered non-inferior if the lower bound of the confidence interval (original scale) is no less than half that of the standard dose, giving a NI margin of 0.5 (NI= -0.301 log10 scale); p = 0.045, t-test, 2 sided — Significance can be considered if P <0.05. Not adjusted for multiple comparisons; Two-sample t-test with unequal variance, noninferiority (NI) margin of 0.5 and two-sided type I error rate of 0.05; Geometric mean titer ratio (GMTR) = 0.7, 95% CI 2-sided [0.5 to 1.0]
Statistical Analysis 2: Comparison: 1 x 10^7 ID MVA-BN vs 1 x 10^8 SC MVA-BN; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.162, t-test, 2 sided — Significance can be considered if P <0.05. Not adjusted for multiple comparisons; Two-sample t-test with unequal variance, noninferiority (NI) margin of 0.5 and two-sided type I error rate of 0.05; Geometric mean titer ratio (GMTR) = 0.4, 95% CI 2-sided [0.3 to 0.6]

2. Secondary Outcome: Individual Peak GMT Through Day 365
Description: Blood was collected at baseline and multiple timepoints post vaccination for evaluation in a vaccinia virus Western Reserve PRNT assay. For each participant, the highest assessment post vaccination was determined as their peak response. For each arm, the geometric mean of peak responses was determined.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 77 | 76
Titer | 215.8 [174.8 to 266.2] | 127.0 [100.1 to 161.1] | 312.0 [238.5 to 408.2]

3. Secondary Outcome: Vaccinia Virus Specific PRNT GMT at Study Day 1, 15, 29, 43, 57, 90, 181, and 365
Description: Blood was collected at baseline and multiple timepoints post vaccination for evaluation in a vaccinia virus Western Reserve PRNT assay. Geometric means were determined for each timepoint.
Time Frame: Day 1 through Day 365
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 77 | 76
Titer
  Day 1 | 10.2 [9.8 to 10.5] | 10.4 [9.8 to 11.1] | 11.2 [9.8 to 12.8]
  Day 15: number analyzed (Participants) | 75 | 76 | 76
  Day 15 | 38.6 [29.9 to 50.0] | 20.8 [16.8 to 25.8] | 39.7 [29.0 to 54.3]
  Day 29: number analyzed (Participants) | 74 | 76 | 76
  Day 29 | 43.7 [33.8 to 56.4] | 24.4 [19.8 to 30.0] | 42.3 [31.0 to 57.6]
  Day 43: number analyzed (Participants) | 74 | 75 | 76
  Day 43 | 203.2 [164.5 to 250.9] | 113.2 [90.3 to 141.9] | 288.9 [222.4 to 375.2]
  Day 57: number analyzed (Participants) | 74 | 76 | 73
  Day 57 | 115.5 [92.2 to 144.7] | 75.6 [61.0 to 93.6] | 175.3 [135.1 to 227.5]
  Day 90: number analyzed (Participants) | 72 | 71 | 72
  Day 90 | 60.2 [48.7 to 74.5] | 36.8 [29.3 to 46.1] | 91.3 [69.0 to 120.8]
  Day 181: number analyzed (Participants) | 74 | 71 | 72
  Day 181 | 25.1 [20.4 to 30.9] | 17.3 [14.2 to 21.1] | 39.7 [28.8 to 54.6]
  Day 365: number analyzed (Participants) | 67 | 66 | 68
  Day 365 | 25.4 [20.2 to 31.9] | 21.7 [16.6 to 28.4] | 41.2 [30.3 to 55.9]

4. Secondary Outcome: Vaccinia Virus Specific PRNT Half-life (t ½)
Description: Half-life, defined as the time from expected peak response (Day 43) to 50% maximal response, was estimated using the first participant visit with titer results less than or equal to half the titer results at Day 43.
Time Frame: Day 43 through Day 365
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 74 | 75 | 75
days | 44 [11 to 326] | 43 [12 to 322] | 43 [9 to 352]
Statistical Analysis 1: Comparison: 2 x 10^7 ID MVA-BN vs 1 x 10^8 SC MVA-BN; Test type: Superiority; p = 0.888, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 1 x 10^7 ID MVA-BN vs 1 x 10^8 SC MVA-BN; Test type: Superiority; p = 0.708, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants Reporting Solicited Systemic AEs Through 14 Days After Each Study Vaccination
Description: Systemic AEs solicited on a memory aid provided to participants included fever, chills, nausea, headache, fatigue, change in appetite, myalgia, and arthralgia. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time through 14 days after each study vaccination (Day 1 through Day 15 for Dose 1 and Day 29-43 for Dose 2).
Time Frame: Day 1 through Day 43
Population: The Safety Analysis population includes all participants who received the first study vaccination. Participants are analyzed according to the study product that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
Participants | 59 | 55 | 62

6. Secondary Outcome: Number of Participants Reporting Solicited Local AEs Through 14 Days After Each Study Vaccination
Description: Local AEs solicited on a memory aid provided to participants included pain at injection site, erythema/redness, induration/swelling (functional grade based on interference with daily activity and any measure value greater than 2.5 cm) and pruritis at injection site. Participants are considered reporting the local AE if they reported mild or greater severity at any time through 14 days after each study vaccination (Day 1 through Day 15 for Dose 1 and Day 29 through 43 for Dose 2).
Time Frame: Day 1 through Day 43
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
Participants | 73 | 75 | 70

7. Secondary Outcome: Number of Participants Reporting Unsolicited Related and Unrelated Adverse Events (AEs) Through 28 Days After Each Vaccination
Description: Frequency of all unsolicited non-serious AEs from day of each study vaccination through 28 days after each vaccination (Day 1 through Day 29 for Dose 1 and Day 29 through Day 57 for Dose 2).
Time Frame: Day 1 through Day 57
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
Participants
  Related AEs | 64 | 62 | 37
  Unrelated AEs | 31 | 26 | 18

8. Secondary Outcome: Number of Participants Reporting Related and Unrelated Medically Attended Adverse Events (MAAEs)
Description: An MAAE is an unsolicited AE that results in unscheduled medical attention such as a hospitalization for less than 24 hours, an emergency room visit, or an otherwise unscheduled healthcare visit for any reason. All MAAEs were collected from Study Day 1 through Study Day 57, and all MAAEs deemed related to the vaccine were collected through Study Day 181.
Time Frame: Day 1 through Day 181
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
Participants
  Related MAAEs | 1 | 0 | 0
  Unrelated MAAEs | 11 | 9 | 4

9. Secondary Outcome: Number of Participants Reporting Related and Unrelated Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. All SAEs were collected from Study Day 1 through Study Day 57, and all SAEs deemed related to the vaccine were collected through Study Day 181.
Time Frame: Day 1 through Day 181
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
Participants
  Related SAEs | 0 | 0 | 0
  Unrelated SAEs | 0 | 1 | 1

10. Secondary Outcome: Number of Participants Who Withdrew or Discontinued Vaccination
Description: Participants could voluntarily withdraw their consent for study participation for any reason at any time. Primary reason for withdrawal was recorded and early termination visits were attempted. Participants who received the first vaccination could choose to discontinue receipt of study vaccine for any reason and could choose to remain in the study (i.e., not withdraw from study). In addition, a participant could be discontinued from receipt of the second vaccination. Discontinuation from vaccination did not mean automatic withdrawal from the study, and participants were monitored for safety and immunogenicity if the participant consented.
Time Frame: Day 1 through Day 365
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
Number analyzed (Participants) | 75 | 78 | 76
participants
  Withdrew | 6 | 9 | 5
  Discontinued Vaccination | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited events, including local and systemic AEs, were collected from the time of each study vaccination through 14 days after each study vaccination. Unsolicited, non-serious AEs, all SAEs, and all MAAEs were collected from the time of first study vaccination through Study Day 57. All related SAEs and MAAEs were collected from the time of each study vaccination through Study Day 181.
Arm/Group | 2 x 10^7 ID MVA-BN | 1 x 10^7 ID MVA-BN | 1 x 10^8 SC MVA-BN
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/78 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/78 | 1/76
Other Adverse Events (participants affected / at risk) | 75/75 | 78/78 | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 x 10^7 ID MVA-BN (N=75) | 1 x 10^7 ID MVA-BN (N=78) | 1 x 10^8 SC MVA-BN (N=76)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 x 10^7 ID MVA-BN (N=75) | 1 x 10^7 ID MVA-BN (N=78) | 1 x 10^8 SC MVA-BN (N=76)
Nausea (Gastrointestinal disorders) | 17 (21) | 15 (18) | 19 (21)
Chills (General disorders) | 15 (15) | 13 (16) | 13 (15)
Fatigue (General disorders) | 43 (60) | 43 (57) | 53 (75)
Injection site discolouration (General disorders) | 58 (94) | 60 (103) | 9 (10)
Injection site exfoliation (General disorders) | 9 (12) | 7 (8) | 0 (0)
Injection site nodule (General disorders) | 51 (68) | 46 (59) | 34 (37)
Injection site erythema (General disorders) | 62 (110) | 56 (89) | 40 (57)
Injection site induration (General disorders) | 68 (154) | 75 (149) | 50 (99) — Functional Grade
Injection site induration (General disorders) | 37 (50) | 33 (39) | 40 (60) — Measurement
Injection site pain (General disorders) | 49 (69) | 44 (64) | 67 (113)
Injection site pruritus (General disorders) | 64 (119) | 73 (125) | 42 (62)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 4 (4)
Appetite disorder (Metabolism and nutrition disorders) | 11 (11) | 17 (21) | 13 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (21) | 12 (14) | 13 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (28) | 19 (25) | 33 (47)
Headache (Nervous system disorders) | 36 (45) | 37 (47) | 43 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT05512949/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT05512949/SAP_002.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT05512949/ICF_000.pdf